CLINICAL TRIAL: NCT03292354
Title: Personalization of CM Injection Protocols in Coronary Computed Tomographic Angiography
Acronym: PeopleCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Joachim Wildberger, Prof.Dr. J.E. Wildberger, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NL59507.068.16
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Coronary Artery Calcification; Cardiac Disease
Keywords: Coronary Computed Tomography Angiography; Image Quality; Contrast Media Reduction; Personalised Injection Protocols
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: All investigators who assess the image quality will be blinded to the assigned contrast media protocol. Only the technicians who complete the scan and injection protocol will be unblinded for the contrast media protocol chosen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Body Weight (BW) (Active Comparator): Patients referred for CCTA in this group receive a personalised contrast media protocol. Contrast media administration based on body weight.
  Interventions: Other: Contrast media administration
- Cardiac output (CO) (Active Comparator): Patients referred for CCTA in this group receive a personalised contrast media protocol. Contrast media administration based on cardiac output.
  Interventions: Other: Contrast media administration
- Lean Body weight (LBW) (Active Comparator): Patients referred for CCTA in this group receive a personalised contrast media protocol. Contrast media administration based on Lean Body Weight.
  Interventions: Other: Contrast media administration
- Control group (No Intervention): Patients in this group will be included retrospectively and have received the standard CM injection protocol previously used in our department.

INTERVENTIONS:
Other: Contrast media administration — All patients will receive contrast media with a concentration of 300 mg I/mL (Iopromide 300). The flowrate and volume will be calculated with help of the different formulas belonging to the three different arms.
  Arms: Body Weight (BW); Cardiac output (CO); Lean Body weight (LBW)

SUMMARY:
Cardiac computed tomography (CCT) is one of the standard non-invasive imaging techniques allowing imaging of the heart and coronary arteries with a high temporal and spatial resolution. The high sensitivity and negative predictive value (NPV) of coronary CT angiography (CCTA) make it a valuable tool in the assessment of coronary artery disease (CAD) in patients with low to intermediate risk for CAD, especially to rule out CAD. This risk stratification can be done with help of multiple different risk-calculators (e.g. the updated Diamond-Forrester model by Genders et al. 2012). These calculators take different variables into account, e.g. advanced age, gender, blood pressure, diabetes mellitus (DM), lipid profile and smoking.

The aim of CCTA is a high diagnostic accuracy, which depends on both optimal intravascular enhancement (in Hounsfield Units; minimal 325 HU) and contrast-to-noise ratio (CNR). Optimal intravascular enhancement and CNR depend on different factors such as scan technique (e.g. tube voltage, tube potential), parameters of the administered contrast material (CM) and patient related factors (e.g. cardiac output (CO), body weight (BW)).

Patients with cardiac diseases often have multiple risk factors for developing contrast induced nephropathy (CIN), e.g. diabetes mellitus, advanced age, hypertension and chronic kidney disease. Although the relationship between CTA and CIN has recently come to discussion (AMACING trial; Nijssen et al. 2017), it is still desirable to minimise the CM volume used in these patients. One method to reduce the CM volume is to personalise the injection protocols. The personalisation of injection protocols to the individual patient is gaining more attention in the field of CT imaging. The goal is to individualise the injection protocols to a level, where the patient only receives the minimal amount of CM needed to acquire a diagnostic scan, while maintaining a diagnostic image quality. Many techniques are available and have been studied, e.g. adjustment of CM volume to scan protocol, CO, lean body weight (LBW) and BW.

However, no data is available on which of these is the most beneficial method for the personalisation of CM injection protocols. Therefore, the aim of this study is to assess the performance of three different personalized injection protocols (based on CO, LBW and BW) in CCTA with regard to image quality in comparison to previously used protocols in our department. We hypothesize that the personalized injection protocols will be non-inferior, provide a homogenous coronary enhancement (less non-diagnostic scans) in patients, and will account for a reduction of CM volume in our department in comparison to the previously used protocols.

DETAILED DESCRIPTION:
Cardiac diseases still are the leading cause of death in the western world. Besides the high mortality of the cardiac disease itself, recent studies have shown an increasing evidence of the prognostic value of cardiac diseases, particularly coronary artery disease (CAD), in a broad variety of other diseases. Especially in patients with oncological pathologies undergoing radiotherapy or lung resection surgery [Ambrogi et al. 2003; Kanzaki et al. 2017; Khakoo et al. 2008; Basacaraju et al. 2002; Fajardo et al. 1972]. Cardiac computed tomography angiography (CCTA) is one of the standard non-invasive imaging techniques allowing imaging of the heart and coronary arteries with a high temporal and spatial resolution. The high sensitivity and negative predictive value (NPV) of CCTA make it a valuable tool in the assessment of CAD. Especially to rule out CAD in patients with low to intermediate risk for CAD [Hendel et al. 2006; Goldstein et al. 2011; Budoff et al. 2008; Meijboom et al. 2008; Roffi et al. 2016].

The aim of CCTA is to achieve a high diagnostic accuracy, which depends on both optimal intravascular enhancement (in Hounsfield Units (HU); minimal 325 HU) and contrast-to-noise ratio (CNR). Optimal intravascular enhancement and CNR depend on multiple factors, such as scan technique (e.g. tube voltage (kV) and tube potential), parameters of the administered contrast material (CM) (e.g. concentration, flow rate) and patient related factors (e.g. body weight (BW), heart rate or cardiac output [CO]) [Bae et al. 2004; Awai et al. 2004]. Dedicated CT protocols are necessary to image the heart and the coronary arteries. These protocols require a correlation to the patient's electrocardiogram (ECG) in order to minimize cardiac motion and deliver a sharp image of the heart and coronary arteries. Depending on the heart rate of the patient, the scan can either be a prospectively ECG-triggered high-pitch or adaptive sequence, or retrospectively ECG-gated helical scan.

Patients with cardiac diseases often have multiple risk factors for developing contrast induced nephropathy (CIN), e.g. diabetes mellitus (DM), advanced age, hypertension, cardiovascular disease and chronic kidney disease. Although the relationship between CTA and CIN has recently come to discussion (AMACING trial; Nijssen et al. 2017), it is still desirable to minimise the CM volume used in these patients. Multiple strategies have been studied to reduce CM volume in CTA imaging [Kok et al 2016; Kok et al. 2015; Kok et al. 2016; Kok et al. 2016, Mihl et al. 2016; Seehofnerova et al. 2015; Hendriks et al. 2016]. For instance, lowering tube voltage to achieve a higher attenuation, the latter explained by the fact that mean photon energy of lower tube voltage settings in the x-ray beam moves closer to the K-edge of iodine (33.2 keV).

The personalisation of injection protocols to the individual patient is gaining more attention in CT imaging, and the goal is to individualise the injection protocols to a level, where the patient only receives the minimal amount of CM needed to make a diagnostic scan with a diagnostic image quality. Besides the techniques mentioned above, other techniques are possible, e.g. adjustment according to patients CO, lean body weight (LBW), and BW.

Both blood volume and CO increase with an increasing BW. When CO increases, the distribution of CM is also increased. On one hand this results in a fastened test bolus arrival, on the other hand in a decreased and shortened intravascular attenuation profile (in comparison to a decreased CO) [Bae KT 2010]. Therefore, both timing and CM volume can be adjusted to CO in order to achieve a similar intravascular attenuation profile.

LBW is a measurement for body fat percentage. It is known that fatty tissue is not as well vascularised in comparison to muscle tissue. Thus with increasing BW due to fatty tissue, the blood volume does not increase linear to BW. For instance, patients with a high BW due to increased muscle tissue, need more CM volume compared to patients with a high BW due to fatty tissue. The concept of LBW accounts for this fact [Bae KT 2010].

When adjusting CM volume to BW, less CM volume is needed with a lower BW in comparison to a higher BW, due to the decreased blood volume and CO [Bae KT 2010].

The tube voltage, set by automated tube voltage selection (ATVS, CAREkV, Siemens, Berlin, Germany), needs to be taken into account as well. CAREkV is a software program which chooses the optimal tube voltage (kV) and tube current (mAs) settings for the individual patient, based on their topograms, while maintaining a diagnostic image quality. Lower kV settings result in a higher intravascular enhancement if the same amount of CM is used, thus giving the potential to decrease CM volume in lower kV settings.

Since no data exist on the optimal method of choice, the aim of this study is to assess the performance of three personalized injection protocols (CO, LBW and BW) in CCTA, in comparison to previously used protocols, with regard to image quality. Secondly we want to assess the presence and severity of CAD in patients undergoing CCTA with help of the coronary artery disease reporting and data system (CAD-RADS).

A total of 330 patients will be included in this prospectively observer blinded randomized controlled non-inferiority trial. All patients will be randomised in one of three groups (CO, LBW and BW) with help of a randomisation software program (ALEA). The control group will consist of 110 consecutive patients who will be included retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for CCTA;
* Age > 18 years;
* Informed consent obtained.

Exclusion Criteria:

* Inability to perform a breath hold for the expected scan time;
* Hemodynamic instability;
* Pregnancy;
* Renal insufficiency (defined as glomerular filtration rate (GFR) < 30 mL/min);
* Iodine allergy;
* Age < 18 years;
* Absence of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Image quality | 1 year
  To evaluate the performance of the individualised injection protocols in CCTA, with regard to intravascular attenuation (minimal 325 HU) and compare them with the control group (non-inferiority).

SECONDARY OUTCOMES:
Objective image quality | 1 year
  The performance of the individualised injection protocols in CCTA with regard to objective image quality (image noise, CNR and SNR as calculated from the intravascular enhancement), compared to the standard injection protocol.
subjective image quality | 1 year
  The performance of the individualised injection protocols in CCTA with regard to subjective image quality (4-point Likert scale), compared to the standard injection protocol.
Coronary artery disease | 1 year
  To assess the presence and severity of coronary artery disease (CAD) with help of the CAD-RADS classification

CONTACTS AND LOCATIONS:
Overall Officials: Joachim E Wildberger, Prof.dr., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Zuid-Limburg, Netherlands

REFERENCES:
- [Background] Ambrogi V, Pompeo E, Elia S, Pistolese GR, Mineo TC. The impact of cardiovascular comorbidity on the outcome of surgery for stage I and II non-small-cell lung cancer. Eur J Cardiothorac Surg. 2003 May;23(5):811-7. doi: 10.1016/s1010-7940(03)00093-9. PMID 12754038
- [Background] Kanzaki R, Inoue M, Minami M, Shintani Y, Funaki S, Kawamura T, Okumura M. Outcomes of lung cancer surgery in patients with coronary artery disease: a decade of experience at a single institution. Surg Today. 2017 Jan;47(1):27-34. doi: 10.1007/s00595-016-1355-z. Epub 2016 May 19. PMID 27194125
- [Background] Khakoo AY, Yeh ET. Therapy insight: Management of cardiovascular disease in patients with cancer and cardiac complications of cancer therapy. Nat Clin Pract Oncol. 2008 Nov;5(11):655-67. doi: 10.1038/ncponc1225. Epub 2008 Sep 16. PMID 18797437
- [Background] Basavaraju SR, Easterly CE. Pathophysiological effects of radiation on atherosclerosis development and progression, and the incidence of cardiovascular complications. Med Phys. 2002 Oct;29(10):2391-403. doi: 10.1118/1.1509442. PMID 12408314
- [Background] Fajardo LF, Stewart JR. Coronary-artery disease after radiation. N Engl J Med. 1972 Jun 8;286(23):1265-6. doi: 10.1056/nejm197206082862315. No abstract available. PMID 5022894
- [Background] Hendel RC, Patel MR, Kramer CM, Poon M, Hendel RC, Carr JC, Gerstad NA, Gillam LD, Hodgson JM, Kim RJ, Kramer CM, Lesser JR, Martin ET, Messer JV, Redberg RF, Rubin GD, Rumsfeld JS, Taylor AJ, Weigold WG, Woodard PK, Brindis RG, Hendel RC, Douglas PS, Peterson ED, Wolk MJ, Allen JM, Patel MR; American College of Cardiology Foundation Quality Strategic Directions Committee Appropriateness Criteria Working Group; American College of Radiology; Society of Cardiovascular Computed Tomography; Society for Cardiovascular Magnetic Resonance; American Society of Nuclear Cardiology; North American Society for Cardiac Imaging; Society for Cardiovascular Angiography and Interventions; Society of Interventional Radiology. ACCF/ACR/SCCT/SCMR/ASNC/NASCI/SCAI/SIR 2006 appropriateness criteria for cardiac computed tomography and cardiac magnetic resonance imaging: a report of the American College of Cardiology Foundation Quality Strategic Directions Committee Appropriateness Criteria Working Group, American College of Radiology, Society of Cardiovascular Computed Tomography, Society for Cardiovascular Magnetic Resonance, American Society of Nuclear Cardiology, North American Society for Cardiac Imaging, Society for Cardiovascular Angiography and Interventions, and Society of Interventional Radiology. J Am Coll Cardiol. 2006 Oct 3;48(7):1475-97. doi: 10.1016/j.jacc.2006.07.003. No abstract available. PMID 17010819
- [Background] Goldstein JA, Chinnaiyan KM, Abidov A, Achenbach S, Berman DS, Hayes SW, Hoffmann U, Lesser JR, Mikati IA, O'Neil BJ, Shaw LJ, Shen MY, Valeti US, Raff GL; CT-STAT Investigators. The CT-STAT (Coronary Computed Tomographic Angiography for Systematic Triage of Acute Chest Pain Patients to Treatment) trial. J Am Coll Cardiol. 2011 Sep 27;58(14):1414-22. doi: 10.1016/j.jacc.2011.03.068. PMID 21939822
- [Background] Budoff MJ, Dowe D, Jollis JG, Gitter M, Sutherland J, Halamert E, Scherer M, Bellinger R, Martin A, Benton R, Delago A, Min JK. Diagnostic performance of 64-multidetector row coronary computed tomographic angiography for evaluation of coronary artery stenosis in individuals without known coronary artery disease: results from the prospective multicenter ACCURACY (Assessment by Coronary Computed Tomographic Angiography of Individuals Undergoing Invasive Coronary Angiography) trial. J Am Coll Cardiol. 2008 Nov 18;52(21):1724-32. doi: 10.1016/j.jacc.2008.07.031. PMID 19007693
- [Background] Meijboom WB, Meijs MF, Schuijf JD, Cramer MJ, Mollet NR, van Mieghem CA, Nieman K, van Werkhoven JM, Pundziute G, Weustink AC, de Vos AM, Pugliese F, Rensing B, Jukema JW, Bax JJ, Prokop M, Doevendans PA, Hunink MG, Krestin GP, de Feyter PJ. Diagnostic accuracy of 64-slice computed tomography coronary angiography: a prospective, multicenter, multivendor study. J Am Coll Cardiol. 2008 Dec 16;52(25):2135-44. doi: 10.1016/j.jacc.2008.08.058. PMID 19095130
- [Background] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S. [2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC)]. G Ital Cardiol (Rome). 2016 Oct;17(10):831-872. doi: 10.1714/2464.25804. No abstract available. Italian. PMID 27869901
- [Background] Bae KT, Tran HQ, Heiken JP. Uniform vascular contrast enhancement and reduced contrast medium volume achieved by using exponentially decelerated contrast material injection method. Radiology. 2004 Jun;231(3):732-6. doi: 10.1148/radiol.2313030497. PMID 15163812
- [Background] Awai K, Hiraishi K, Hori S. Effect of contrast material injection duration and rate on aortic peak time and peak enhancement at dynamic CT involving injection protocol with dose tailored to patient weight. Radiology. 2004 Jan;230(1):142-50. doi: 10.1148/radiol.2301021008. PMID 14695390
- [Background] Kok M, Mihl C, Hendriks BM, Altintas S, Kietselaer BL, Wildberger JE, Das M. Optimizing contrast media application in coronary CT angiography at lower tube voltage: Evaluation in a circulation phantom and sixty patients. Eur J Radiol. 2016 Jun;85(6):1068-74. doi: 10.1016/j.ejrad.2016.03.022. Epub 2016 Mar 22. PMID 27161054
- [Background] Kok M, Mihl C, Seehofnerova A, Turek J, Jost G, Pietsch H, Haberland U, Wildberger JE, Das M. Automated Tube Voltage Selection for Radiation Dose Reduction in CT Angiography Using Different Contrast Media Concentrations and a Constant Iodine Delivery Rate. AJR Am J Roentgenol. 2015 Dec;205(6):1332-8. doi: 10.2214/AJR.14.13957. PMID 26587942
- [Background] Kok M, de Haan MW, Mihl C, Eijsvoogel NG, Hendriks BM, Sailer AM, Derks K, Schnerr RS, Schurink GW, Wildberger JE, Das M. Individualized CT Angiography Protocols for the Evaluation of the Aorta: A Feasibility Study. J Vasc Interv Radiol. 2016 Apr;27(4):531-8. doi: 10.1016/j.jvir.2016.01.009. Epub 2016 Mar 2. PMID 26948327
- [Background] Kok M, Turek J, Mihl C, Reinartz SD, Gohmann RF, Nijssen EC, Kats S, van Ommen VG, Kietselaer BL, Wildberger JE, Das M. Low contrast media volume in pre-TAVI CT examinations. Eur Radiol. 2016 Aug;26(8):2426-35. doi: 10.1007/s00330-015-4080-x. Epub 2015 Nov 11. PMID 26560728
- [Background] Mihl C, Kok M, Altintas S, Kietselaer BL, Turek J, Wildberger JE, Das M. Evaluation of individually body weight adapted contrast media injection in coronary CT-angiography. Eur J Radiol. 2016 Apr;85(4):830-6. doi: 10.1016/j.ejrad.2015.12.031. Epub 2016 Jan 7. PMID 26971431
- [Background] Seehofnerova A, Kok M, Mihl C, Douwes D, Sailer A, Nijssen E, de Haan MJ, Wildberger JE, Das M. Feasibility of low contrast media volume in CT angiography of the aorta. Eur J Radiol Open. 2015 Apr 28;2:58-65. doi: 10.1016/j.ejro.2015.03.001. eCollection 2015. PMID 26937437
- [Background] Hendriks BM, Kok M, Mihl C, Bekkers SC, Wildberger JE, Das M. Individually tailored contrast enhancement in CT pulmonary angiography. Br J Radiol. 2016;89(1061):20150850. doi: 10.1259/bjr.20150850. Epub 2016 Jan 22. PMID 26689096
- [Background] Bae KT. Intravenous contrast medium administration and scan timing at CT: considerations and approaches. Radiology. 2010 Jul;256(1):32-61. doi: 10.1148/radiol.10090908. PMID 20574084
- [Background] Genders TS, Steyerberg EW, Hunink MG, Nieman K, Galema TW, Mollet NR, de Feyter PJ, Krestin GP, Alkadhi H, Leschka S, Desbiolles L, Meijs MF, Cramer MJ, Knuuti J, Kajander S, Bogaert J, Goetschalckx K, Cademartiri F, Maffei E, Martini C, Seitun S, Aldrovandi A, Wildermuth S, Stinn B, Fornaro J, Feuchtner G, De Zordo T, Auer T, Plank F, Friedrich G, Pugliese F, Petersen SE, Davies LC, Schoepf UJ, Rowe GW, van Mieghem CA, van Driessche L, Sinitsyn V, Gopalan D, Nikolaou K, Bamberg F, Cury RC, Battle J, Maurovich-Horvat P, Bartykowszki A, Merkely B, Becker D, Hadamitzky M, Hausleiter J, Dewey M, Zimmermann E, Laule M. Prediction model to estimate presence of coronary artery disease: retrospective pooled analysis of existing cohorts. BMJ. 2012 Jun 12;344:e3485. doi: 10.1136/bmj.e3485. PMID 22692650
- [Background] Nijssen EC, Rennenberg RJ, Nelemans PJ, Essers BA, Janssen MM, Vermeeren MA, Ommen VV, Wildberger JE. Prophylactic hydration to protect renal function from intravascular iodinated contrast material in patients at high risk of contrast-induced nephropathy (AMACING): a prospective, randomised, phase 3, controlled, open-label, non-inferiority trial. Lancet. 2017 Apr 1;389(10076):1312-1322. doi: 10.1016/S0140-6736(17)30057-0. Epub 2017 Feb 21. PMID 28233565